CLINICAL TRIAL: NCT00823498
Title: Perceptions of School, Recreation, and Transportation Environments Among African American Families in Public Housing--II
Brief Title: Physical Activity in Public Housing - II
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0610
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: Cancer Prevention; African American; African American Parents; African American Youth; Public Housing; Physical Activity; Focus Groups; Housing Developments; Houston Public Housing; Photovoice Project; Prevention
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Focus Groups; Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African American Parents
  Interventions: Behavioral: Interview; Other: Photovoice Project
- African American Youth: African American Youth between ages of 12-15 Years Old
  Interventions: Behavioral: Focus Group; Behavioral: Interview; Other: Photovoice Project

INTERVENTIONS:
Behavioral: Focus Group — 6 Focus Groups asked how living in public housing effects physical activity and feelings about neighborhood.
  Groups: African American Youth
Behavioral: Interview — Interview with a member of study staff at housing development site.
  Other Names: Survey
Other: Photovoice Project — Activity allowing expression of thoughts and feelings about neighborhood through neighborhood pictures taken by youth and parent(s).

SUMMARY:
The aims of the proposed study are to:

1. Examine how youth and their parents use and perceive three active living domains for physical activity (PA): schools, recreation, and transportation environment;
2. Identify patterns and predictors of environmental perceptions of physical activity;
3. Compare and contrast youth evaluations of physical activity resources with research team objective evaluations of physical activity resources;
4. Using above data, refine the conceptual framework of physical activity phenomena in low-income minority communities guiding this research and develop items for a quantitative survey measuring parental and youth environmental perceptions of physical activity for a future trial with this population.

DETAILED DESCRIPTION:
Cognitive Interview:

If you agree to take part in this study, you will have an interview to discuss the questions asked in the a physical activity survey. You will read the survey and be asked about what you thought when you read certain questions and how well you understood the questions.

The interview will be recorded with a tape recorder and the results will be written down. Your name will not be used during the interview and will not be recorded. You will only be identified by a number given to you by the study staff. After the interview comments are written down, the interview tape will be destroyed. The transcript will be stored in a safe locked compartment for 3 years, then it will be destroyed.

Length of Study:

You will be off study after the interview.

THIS IS AN INVESTIGATIONAL STUDY.

Up to 8 children and 4 parents will take part in this study. All will be enrolled at M. D. Anderson.

Physical Activity in Public Housing II -- Parent:

If you agree to take part in this study, you will take part in an interview with a member of the study staff at your housing development site. During the interview, you will be asked if living in public housing has any effect on your options for physical activity and how you feel about your neighborhood. The interview will take about 45 minutes to complete.

The interview will be recorded with a tape recorder and the results will be written down. Your name will not be used during the interview and will not be recorded. You will only be identified by a number given to you by the study staff. After the interview comments are written down, the interview tape will be destroyed. The transcript will be stored in a safe locked compartment for 3 years, then it will be destroyed.

At the time of the interview, you will also be given a survey that will have questions about how you feel about your neighborhood, access to recreational facilities, physical activity, how the people around you feel about exercise, and sociodemographic information (such as age and sex). The survey will take about 20 minutes to complete.

Photovoice Project:

You may be randomly selected (as in the flip of a coin) to receive a letter asking you to participate in the Photovoice project. The Photovoice project is an activity that will allow you to express your thoughts and feelings about your neighborhood through pictures that you and your child will take of your neighborhood. You and your child will take pictures of your neighborhood with a camera provided to you by the study staff. The pictures will be developed by the study staff and they will bring them back to your house. You and your child will then participate in an interview to talk about the photographs you took. This interview will take about 20 minutes.

Length of Study:

If you are selected and choose to take part in the Photovoice project, you will be off study after the Photovoice interview. If you do not chose to take part in the Photovoice project, you will be off study after the survey.

THIS IS AN INVESTIGATIONAL STUDY.

Up to 36 adult parents will take part in an individual interview. In total 36 parents and 36 youth will take part in this study for a total of 72 participants. All will be enrolled at M. D. Anderson.

Physical Activity in Public Housing II -- Youth:

If you agree to take part in this study, you will take part in a focus group. A focus group is a group of people who are asked questions about certain topics and then discuss these topics with other group members. During the focus group, you will talk about how living in public housing effects your physical activity and how you feel about your neighborhood. There will be 6 focus groups, each made up of 6 participants. The focus group session will take about 45 minutes.

The focus group session will be recorded with a tape recorder and the results will be written down. Your name will not be used during the interview and will not be recorded. You will only be identified by a number given to you by the study staff. After the interview comments are written down, the interview tape will be destroyed. The transcript will be stored in a safe locked compartment for 3 years, then it will be destroyed.

At the time of the focus group session, you will also be given a survey that will have questions about how you feel about your neighborhood, access to recreational facilities, physical activity, and how the people around you feel about exercise. The survey will take about 15 minutes to complete.

Photovoice Project:

You may be randomly selected (as in the flip of a coin) to receive a letter asking you to participate in the Photovoice project. The Photovoice project is an activity that will allow you to express your thoughts and feelings about your neighborhood through pictures that you and your parent will take of your neighborhood. You and your parent will take pictures of your neighborhood with a camera provided to you by the study staff. The pictures will be developed by the study staff and they will bring them back to your house. You and your parent will then participate in an interview to talk about the photographs you took. This interview will take about 20 minutes.

Length of Study:

If you are selected and choose to take part in the Photovoice project, you will be off study after the Photovoice interview. If you do not chose to take part in the Photovoice project, you will be off study after the survey.

THIS IS AN INVESTIGATIONAL STUDY.

Up to 36 youth will take part in a focus group. In total 36 parents and 36 youth will take part in this study for a total of 72 participants. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Being able to read and speak English
2. Self-identify as African American or black
3. Youth between the ages of 12-15 years old
4. Adults must be the biological parent or legal guardian of the participating child
5. Youth and parents must live in the housing development at least 50% of the time
6. Adults must have a child who also is participating in the study
7. Children must have a parent or legal guardian who also is participating in the study

Exclusion Criteria:

1) None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: African American parents and youth residing in selected Houston public housing developments.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2009-01-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Parent/Child Perceptions of School, Recreational, + Transportation Environments among African American youth in Public Housing | 2 Years; Qualitative + Quantitative Data from In-depth Interviews and Focus Groups

SECONDARY OUTCOMES:
Effects of public housing on physical activity. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H McNeill, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org